CLINICAL TRIAL: NCT00271440
Title: Effect of Chlorhexidine Cleansing on Skin Flora of Newborns in Nepal
Acronym: NNIPS-SFS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Tribhuvan University, Nepal (Other); Nepal Nutrition Intervention Project Sarlahi (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01-HD44004-2; R01HD044004 (NIH)
Record Dates: First submitted 2005-12-29; First posted 2006-01-02 (Estimated); Last update posted 2010-04-05 (Estimated); Status verified 2010-04

CONDITIONS: Bacterial Infection
Keywords: chlorhexidine; neonatal; skin flora; skin cleansing; bacterial colonization
MeSH Terms: conditions — Bacterial Infections | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CHX 1.0% (Experimental): 1.0% CHX wiping
  Interventions: Procedure: skin cleansing with chlorhexidine (0.25%, 0.5%, 1%)
- CHX 0.5% (Experimental): 0.5% Chlorhexidine
  Interventions: Procedure: skin cleansing with chlorhexidine (0.25%, 0.5%, 1%)
- CHX 0.25% (Experimental): chlorhexidine cleansing with pre-soaked pre-sealed wipe
  Interventions: Procedure: skin cleansing with chlorhexidine (0.25%, 0.5%, 1%)

INTERVENTIONS:
Procedure: skin cleansing with chlorhexidine (0.25%, 0.5%, 1%)

SUMMARY:
The purpose of this study is to compare the reductions in skin flora of newborns after a single cleansing of the body with three concentrations of chlorhexidine (0.25%, 0.5%, 1.0%) and to examine the safety of skin cleansing in neonates in Nepal.

DETAILED DESCRIPTION:
Studies in Malawi, Egypt, and Nepal suggest that neonatal skin cleansing with chlorhexidine solutions may reduce the risk of infection and mortality. Cleansing with 0.25% chlorhexidine in Nepal resulted in a 28% reduction in mortality among low birth weight infants, while there was no impact on infants of normal weight. The mechanism of action for this observed benefit is not clear. Chlorhexidine may remove pathogens from the skin of the newborn and/or prevent exposure to pathogens that may otherwise cause infection and lead to sepsis. The benefit of chlorhexidine cleansing may be extended with higher concentrations of chlorhexidine.

Infants born at the Tribhuvan University Teaching Hospital in Katmandu, Nepal will be randomized to skin cleansing with chlorhexidine at one of three concentrations (0.25%, 0.50%, 1.00%). Skin swabs will be collected before wiping, and two and twenty-four hours after wiping in order to compare levels of bacteria on the skin across the treatment groups. A small quantity of blood will be collected at 24 hours after wiping to determine the potential for absorption of chlorhexidine

ELIGIBILITY:
Inclusion Criteria:

* babies born at Tribhuvan University Teaching Hospital
* greater than 1500 grams

Exclusion Criteria:

* less than 1500 grams
* requires major surgical procedure
* clinically evident skin infection
* generalized skin disease
* major congenital anomoly

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 286 (Actual)
Dates: Start 2006-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Skin flora reduction across treatment groups | prior to wipe, 2hrs after, and 24hrs after

SECONDARY OUTCOMES:
Serum concentrations of chlorhexidine 24 hours after wipe | 24 hrs after wipe

CONTACTS AND LOCATIONS:
Overall Officials: Luke C Mullany, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Tribhuvan University Teaching Hospital, Kathmandu, Nepal